CLINICAL TRIAL: NCT02068703
Title: Use of Sleep Enhancing Tools Impact on Self-Reported Sleep Survey
Brief Title: Sleep Enhancing Tools: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Peter Farrehi MD, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00075628
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Sleep; Pain
Keywords: survey
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Subjects will receive a 10 minute presentation, aimed at educating on the value of sleep PLUS a demonstration of tools (face mask, ear plugs and white noise machine) to improve sleep.
  Interventions: Behavioral: Sleep Education Presentation; Behavioral: Sleep Tool Demonstration
- Inert Control (Placebo Comparator): Same 10 min time exposure and tool delivery to subjects in this arm WITHOUT demonstration.
  Interventions: Behavioral: Sleep Education Presentation

INTERVENTIONS:
Behavioral: Sleep Education Presentation — Subjects will receive a 10 minute presentation, aimed at educating on the value of sleep WITHOUT a demonstration of tools to improve sleep.
Behavioral: Sleep Tool Demonstration — Subjects will receive a 10 minute presentation, aimed at educating on the value of sleep PLUS a demonstration of tools to improve sleep.
  Arms: Intervention

SUMMARY:
To demonstrate whether use of sleep enhancing aids (face mask, ear plugs or white noise machine) in hospitalized patients can positively affect subjective symptoms of sleep quality, fatigue and pain.

DETAILED DESCRIPTION:
A randomized, clinical pilot to trial the effect of sleep tools on patients' perception of sleep within the hospital setting.

We propose to conduct this pilot study to improve subjective symptoms of sleep deprivation in non-ICU hospitalized subjects by performing a brief intervention, easily performed at the point of care. Given the heterogeneity of hospitalized patients with varying ages, co-morbidities and other factors (such as pain and fatigue), we felt that an initial pilot study should focus on acceptability of three sleep aids (ear plugs, eye masks and white noise machine) among hospitalized non-ICU patients. Patients will be able to choose which aid they use and will be allowed to change aids during their hospital stay.

The primary outcomes of this study will be 1) improvement in perceived sleep quality as measured by PROMIS, a validated patient-reported outcome information system and 2) quality of care measures (length of stay, medication use and participation in therapy sessions).

PROMIS (Patient Reported Outcomes Measurement Information System) is an NIH sponsored health survey tool.

Information on characteristics (both patient and environment) including demographics, illness severity, number of medications, specific medications (such as sedatives and pain medications) will be collected to examine which predictors of improved perception of sleep quality correlate with use of sleep aids. This study is intended to focus on modifying the environment at the patient level rather than addressing the sources of environmental hospital noise.

Our study has the potential to impact this field with a preventative education based intervention, using simple tools in the non-ICU setting. It is important to understand this is not a study measuring sleep objectively but whether hospitalized patients perceive they sleep better if sleep aids are used.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a private room in the hospital
* Speak and read english
* expected length of stay > 2 days

Exclusion Criteria:

* Hearing aids
* sleep apnea using positive airway pressure therapy
* medically or behaviorally unstable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Aggregate change in sleep /pain / fatigue scores on Patient Reported Outcomes Measurement Information System (PROMIS) survey sampled in hospital from baseline to day 3 between study groups | Baseline to day 3
  Change from baseline in sleep / pain / fatigue scores on PROMIS survey in the hospital. Each score ranges from 1-5, 1 equals not at all; 5 equals Very much.

SECONDARY OUTCOMES:
Effect of use of sleep tool devices on length of stay | number hospital days between administration of tool and hospital discharge
  Whether the intervention of demonstrating use of sleep enhancing tools will translate into reduced length of hospital stay

OTHER OUTCOMES:
Effect of sleep enhancing tools on medication use | baseline to day 3
  Whether the intervention of demonstrating use of sleep enhancing tools will translate into reduced use of sleep or pain medication
Effect of sleep enhancing tools on participation in Occupational therapy | baseline to day 3
  Whether the intervention of using sleep enhancing tools will translate into increased number of days participating in therapy during the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Farrehi, MD, Principal Investigator — University of Michigan
Locations (1):
- UMichigan, Ann Arbor, Michigan, United States